CLINICAL TRIAL: NCT00486096
Title: Femoral Arterial Cannulation in Infants Following Complicated Sternal Re-entry
Brief Title: Femoral Arterial Cannulation
Status: Terminated | Type: Observational
Why Stopped: sufficient data collected.
Sponsor: Children's Healthcare of Atlanta (Other)
Other Study IDs: 07-012
Record Dates: First submitted 2007-06-12; First posted 2007-06-13 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2007-06

CONDITIONS: Congenital Disorders
Keywords: cannulation; infant; femoral arterial
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Many children undergoing surgery for congenital heart disease have had prior operations. Re-operative sternotomy carries with it the risk of cardiac injury and the need for emergent peripheral cannulation.

Our first aim is to demonstrate that peripheral arterial cannulation may be lifesaving in cases of complicated sternal re-entry in children and that angio-catheters can be utilized when vessels are too small for standard cannulas.

Our secondary aim is to present a case report of successful femoral cannulation in a 5 kg child.

DETAILED DESCRIPTION:
In children, many of the standard operative sites are either occluded, stenosed, or too small for the smallest manufactured cannulas. In these instances, it may be feasible to utilize angio-catheters for arterial access until central cannulation can be achieved safely. In an in vitro model, we have simulated a cardiopulmonary bypass circuit and arterial cannulation with angio-catheters.

It appears that angio-catheters may be used with acceptable flow hemodynamics for blood vessels too small for standard cannulas.

We have performed this successfully in a 5 kg child.

We have completed the cardiopulmonary bypass model and are ready to submit the hemodynamic data. We would like to submit to a national meeting and hopefully for publication thereafter.

ELIGIBILITY:
Inclusion Criteria:

* case report of successful angio-catheter use on 5 kg child

Exclusion Criteria:

* that which does not meet inclusion criteria

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric children of successful angio-catheter use on 5 kg child
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2007-02; Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian E Kogon, MD, Principal Investigator — Emory Univ. / Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States